CLINICAL TRIAL: NCT02819830
Title: A Randomised Controlled Trial Assessing the Effects of a Six-week Exercise Programme on Fitness, Inflammation and Cardiovascular Risk in Women With Rheumatoid Arthritis
Brief Title: The Effects of a Six-week Exercise Programme Undertaken by Women With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siobhan Graham (Other)
Collaborators: University of Bath (Other)
Responsible Party: Sponsor-Investigator, Siobhan Graham, General Practitioner, Belfast Health and Social Care Trust
Organization: Belfast Health and Social Care Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC: 16/SS/0064
Record Dates: First submitted 2016-06-25; First posted 2016-06-30 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis; Physical Activity
Keywords: Aerobic exercise; Strength training; Inflammation; cardiovascular disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Participants, who have been randomly assigned to the intervention group, will take part in a six-week supervised exercise training programme. This programme takes place in a rehabilitation gymnasium. The exercise programme consists of two group sessions per week (scheduled for evenings, after typical working hours, approximately 12 patients per session). Each session lasts for approximately 70 minutes and includes a 5 minute warm up, 30 minutes of aerobic cycling exercise, 30 minutes of strength training, and a 5 minute cool down.
  Participants will also perform a 30 minute walk each weekend as part of the intervention.
  Interventions: Behavioral: Exercise Intervention
- Control group (No Intervention): Participants who have been randomly assigned to the control group will not undertake the exercise intervention. These participants are instructed to maintain their usual lifestyle.

INTERVENTIONS:
Behavioral: Exercise Intervention — Combined strength and aerobic exercise
  Arms: Intervention group

SUMMARY:
This study is investigating whether a six-week exercise training programme, designed for patients with Rheumatoid Arthritis, improves disease activity, inflammation, cardiorespiratory fitness, muscle strength, flexibility and risk factors for cardiovascular disease. Twenty four patients will be randomly assigned to an intervention or control group (n=12 in each group). The intervention group will will undertake a fully supervised structured exercise training programme, consisting of both aerobic and strength training exercise, taking the form of two 70-minute group fitness classes per week for six weeks. These participants will also undertake a 30-minute walk in their own time. The control group will continue to go about their normal daily activities. Measurements will be made before and after the intervention/control period, including assessments of disease activity (e.g., by gauging how swollen and tender patients' joints are using the Disease Activity Score(DAS) ) and assessments of fitness and/or physical functioning (e.g., 200 meter timed walk test, a strength test, a flexibility test, Health Assessment Questionnaire Disability Index (HAQDI)). Blood samples will also be collected from patients before and after the intervention/control period to measure markers of inflammation, such as C-reactive protein (CRP) and Erythrocyte Sedimentation Rate (ESR). The investigators will also measure other parameters that are linked to type II diabetes (e.g., fasting glucose concentration) and factors implicated in cardiovascular disease risk (e.g., lipid profile and resting blood pressure).

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a multi-system autoimmune disease characterised by chronic inflammation (i.e., a persistent and inappropriate immune response). It primarily affects the joints, causing swelling, pain, reduced muscle strength and high biomarkers of inflammation such as C-Reactive Protein (CRP) and Erythrocyte Sedimentation Rate (ESR). This immune response also results in accelerated atherosclerotic processes, decreased Bone Mineral Density (BMD) and damage to cartilage in the affected joints. Until the mid-1990s, patients with RA had traditionally been advised to avoid physical exercise, due to concerns it may result in progression of joint damage; hospital admission for bed rest was common practice. However, in the last 20 years, studies have shown that combined moderate-intensity aerobic exercise and strength training, can improve joint swelling, increase cardiorespiratory fitness and strength, without exacerbating pain or joint damage in patients with RA. Thus, the American College of Sports Medicine (ACSM) recommends that patients with RA walk or cycle for at least 30 minutes three times a week at a moderate intensity of 60% to 85% of maximum heart rate (HRmax) to improve cardiorespiratory fitness. The ACSM also recommends static or dynamic strength training of all large muscle groups twice weekly, performing three sets of 8-10 repetitions of 50% to 80% of one repetition maximum (1RM). While it is now established that exercise training can limit disease activity, and lower systemic inflammation, it is unclear whether short (e.g., six-weeks) and feasible exercise training programmes (e.g., two 70 minute sessions per week) elicit the same effects as the commonly employed interventions that are more demanding (e.g., 3-12 months; 3-5 sessions per week). In addition, it is unclear whether such a short intervention can modify other factors implicated in non-communicable disease, such as type II diabetes and cardiovascular risk (e.g., glucose control, lipid profile, blood pressure).

Objectives:

To examine if a six-week moderate intensity aerobic exercise and muscle strengthening programme:

* Results in changes in disease activity.
* Improves cardiorespiratory fitness, strength and flexibility.
* Reduces disease related inflammatory markers.
* Reduces blood pressure, improves lipid profile and improves glucose control.

Study Design:

Twenty-four patients will be randomised to either the exercise intervention (n= 12) or the control group (n = 12). The exercise intervention will consist of combined aerobic and strength training group-exercise intervention lasting six weeks, with two classes per week. All participants will undergo assessments to measure markers of inflammation, disease activity, physical fitness, strength, flexibility and cardiovascular risk factors before and after the six-week intervention.

Recruitment:

Female patients aged 18 to 69 years of age with RA attending Rheumatology outpatient clinics at the Belfast and Social Health Care Trust hospitals will be invited to participate. Patients satisfying the inclusion and exclusion criteria who would like to take part will attend two appointments before being randomised to either the six-week exercise intervention or the control group. Following the six-week intervention all patients will return for two further appointments to repeat all measurements taken before the intervention.

Measurements before the six-week intervention.

* Experimental Visit One. This visit is scheduled between 08:00-09:00 (duration 1 hour). Following written consent blood samples, blood pressure, anthropometry, joint examination, questionnaires will be carried out. All patients, in both groups, will be advised to arrive fasted with their last meal to have been eaten greater than 12 hours before arrival. Patients should refrain from exercise during the 48 hours before, and abstain from alcohol and caffeine for 24 hours.
* Experimental Visit Two. This visit is scheduled between 12:00-16:00 (duration 1 hour) and will consist of a 200 metre walk test, a sit and reach flexibility test, and strength test.

Measurements after the six-week intervention:

* Experimental Visit Three. This visit is scheduled between 08:00-09:00 (duration 1 hour). It is identical to visit one. Measurements include a blood sample, blood pressure, anthropometry, joint examination, questionnaires. All participants in both groups will be advised to arrive fasted with their last meal to have been eaten at least 12 hours before arrival. Patients should refrain from exercise during the 48 hours before, and abstain from alcohol and caffeine for 24 hours.
* Experimental Visit Four. This visit is scheduled between 12:00-16:00 (duration 1 hour) it is identical to visit two and consists of the 200 metre walk test, a sit and reach flexibility test, and strength test.

Exercise Intervention:

The six-week exercise programme will comprise two 70-minute group exercise classes per week (usually 12 patients per class). Classes will be fully supervised and will be conducted at a fitness and rehabilitation gymnasium. Each class will consist of four parts (A-D, see below). Participants will also be asked to go for a moderate intensity walk once a week for 30 minutes and maintain an exercise diary for all exercises including gym sessions.

A. Warm up and stretching for five minutes:

The warm-up will begin with standing and raising knees alternately for 30 seconds followed by gentle stretching of all the large muscles groups: lumbar, quadriceps, hamstrings, groin, pectorals, triceps, biceps, hands and feet muscles; stretching of each group will last for 30 seconds. Stretches will be modified for each patient and supportive props used where necessary.

B. Aerobic exercise for 30 minutes:

Aerobic exercise will consist of 30 minutes cycling on a stationary cycle ergometer. This will begin with a five-minute, low-intensity warm-up (low intensity is Heart Rate(HR) < 50% of age predicted HRmaximum). Intensity will then increase to 60% HRmax for 20 minutes, ending with a five-minute low intensity cool-down.

The exercise programme will be progressive, each week increasing in intensity by 5% of HRmax up to 85% HRmax during the final week. Patients will wear a wrist and chest heart-rate monitor, and will be advised when they have reached required intensity. This will be recorded at each class in their exercise diary along with minutes cycled. Progression of intensity will begin after week two to allow for familiarisation with the programme.

C. Strengthening exercises for 30 minutes:

This will consist of five exercises, working the large muscles of the upper limbs, lower limbs and abdomen: leg extension, bench press, low row, modified abdominal crunch and wall squat. Leg extension and low row will be performed on a pulley weights machine and bench press using the multi-gym system.

One repetition maximum (RM) is the maximum weight in kilograms that can be lifted once and no more. Each of these exercises will start with three sets of 8-10 repetitions at 60% of 1RM, progressing by 5% of 1RM each week. RM will be recalculated weekly after week two. Modified abdominal crunch will begin by assessing the maximum number of crunches the patient can perform to near exhaustion. The participants will then perform this number two more times with a 90 second rest in between. After two weeks this will be progressed by recalculating the number of crunches to near exhaustion each week.

The wall squat will start with assessment of the time the patient can hold the squat before becoming fatigued. This will be repeated twice more, with a 90 second rest in between. After two weeks this will be progressed by re-timing the wall squat until fatigue, each week thereafter.

A record of all exercises performed, along with weights lifted, times, and heart rate will be documented weekly by each patient in their record sheets.

D. Cool-down:

Five minutes of light stretching of all the large muscle groups and instructions on performing moderate intensity walk each weekend. The cooI-down is identical to the warm-up.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-69
* Non-smokers
* Diagnosis of Rheumatoid Arthritis for greater than 12 months
* Stable Disease modifying medication for the preceding three months
* Functional capacity class I-II
* Able to use an exercise bicycle
* Willing to exercise twice-weekly on a fixed schedule
* Available for eight weeks between May and September 2016

Exclusion Criteria:

* Cardiovascular disease (i.e. coronary heart disease, previous heart attack, angina, stroke or uncontrolled hypertension)
* Major psychiatric illness, such as schizophrenia or major depression
* A prosthetic hip or knee joint.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in DAS (Disease Activity Score) | Before and after six-week intervention (approximately 8 weeks)
  DAS-28 uses the number of swollen joints, the number of tender joints, the C-reactive Protein level and the patient's global assessment of well-being, scored out of 100, to calculate the disease activity score at that point in time. Based on the American college of rheumatology (ACR) a change of minus 20 % the DAS-28 score is considered a moderate response.
200m Walk-test to estimate Cardiorespiratory fitness | Before and after six-week intervention (approximately 8 weeks)
  Time taken to complete the 200 metre walk test before and after six-week intervention. Measured in seconds.
Strength of quadriceps muscles | Before and after six-week intervention(approximately 8 weeks)
  Using a Cybex dynamometer the investigators will measure the peak muscle torque of a concentric contraction of the quadriceps muscle. This is measured in Newtons metres (N. m)
Flexibility of hamstring muscles | Before and after six-week intervention (approximately 8 weeks)
  Assessed using the Sit and Reach Test box. The patient is seated with feet flat against the sit and reach box. The patient then reaches their arms forward toward the top of the box which has a scale starting at zero centimetres at the participant's ankle up to 40 centimetres beyond the participant's ankle. Increased measurement corresponds to increased hamstring flexibility. Three attempts are recorded and the average measurement in centimetres is recorded. This estimates flexibility of hamstring muscles.
Strength of hamstring muscles | Before and after six-week intervention(approximately 8 weeks)
  Using the Cybex dynamometer the investigators will measure the peak muscle torque of a concentric contraction of the hamstring muscles. This is measured in Newtons metres.
Blood pressure | Before and after six-week intervention (approximately 8 weeks)
  Measured on the left arm of the patient using a sphygmomanometer. The patient will be seated for at least 15 minutes with the arm supported at the level of the precordium. Three measurements will be made and the average recorded in millimetres of mercury (mmHg)
Cardiovascular Risk Score | Before and after six-week intervention (approximately 8 weeks)
  This is calculated using an algorithm call the Q-Risk2 which is validated for use in the United Kingdom. It uses blood pressure, cholesterol level, smoking status, age, body mass index,ethnicity, and presence of rheumatoid Arthritis, chronic kidney disease and family history of heart disease, to predict the ten year risk of cardiovascular disease

SECONDARY OUTCOMES:
CRP (C-Reactive Protein) | Before and after six-week intervention (approximately 8 weeks)
  Marker of inflammation assessed in serum. Measured in milligrams per litre (mg/litre)
ESR (Erythrocyte Sedimentation Rate) | Before and after six-week intervention (approximately 8 weeks)
  Marker of inflammation. Units of measurement are millimetres per hour (mm/hour)
BMI (Body Mass Index) | Before and after six-week intervention (approximately 8 weeks)
  The investigators will firstly measure the patient's weight in kilograms and the participant's height in metres. BMI is calculated by dividing the participant's weight by the participant's height squared. Units of measurement are kilograms per metre squared (kg/ m2)
Fasting glucose | Before and after six-week intervention (approximately 8 weeks)
  Assessed after 12 hours fasting. Units of measurement are millimoles per litre (mmol/L)
HBA1C (Glycated Haemoglobin 1C) | Before and after six-week intervention(approximately 8 weeks)
  Assessed 12 hours after fasting. Units of measurement are millimoles per mole (mmol/mol)
Fasting total cholesterol | Before and after six-week intervention (approximately 8 weeks)
  Assessed 12 hours after fasting. Measured in millimoles per litre (mmol/L)
Fasting HDL-Cholesterol | Before and after six-week intervention (approximately 8 weeks)
  Assessed 12 hours after fasting. Measured in millimoles per litre (mmol/L)
Fasting LDL-Cholesterol | Before and after six-week intervention (approximately 8 weeks)
  Assessed 12 hours after fasting. Measured in millimoles per litre (mmol/L)
Fasting Triglycerides | Before and after six-week intervention (approximately 8 weeks)
  Assessed 12 hours after fasting. Measured in millimoles per litre (mmol/L)
HAQDI (Health Assessment Questionnaire Disability Index) | Before and after six-week intervention (approximately 8 weeks)
  Qualitative assessment of functional capacity to assess ability to carry out activities of daily living
The short form of the International Physical Activity Questionnaire (IPAQ) | Before and after six-week intervention (approximately 8 weeks)
  An assessment of the type and quantity in hours and minutes of physical activity during the previous week.

CONTACTS AND LOCATIONS:
Overall Officials: James E Turner, BSc PhD, Principal Investigator — University of Bath; Claire Riddell, MD MB BCH, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Musgrave Park Hospital, Belfast health and social care trust., Belfast, County Down, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] ACSM 2010. American College of Sports Medicine's Resource Manual for Guidelines for Exercise Testing and Prescription. 6th Edition, 659-661.
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Crowson CS, Liao KP, Davis JM 3rd, Solomon DH, Matteson EL, Knutson KL, Hlatky MA, Gabriel SE. Rheumatoid arthritis and cardiovascular disease. Am Heart J. 2013 Oct;166(4):622-628.e1. doi: 10.1016/j.ahj.2013.07.010. Epub 2013 Aug 29. PMID 24093840
- [Background] de Jong Z, Munneke M, Kroon HM, van Schaardenburg D, Dijkmans BA, Hazes JM, Vliet Vlieland TP. Long-term follow-up of a high-intensity exercise program in patients with rheumatoid arthritis. Clin Rheumatol. 2009 Jun;28(6):663-71. doi: 10.1007/s10067-009-1125-z. Epub 2009 Feb 27. PMID 19247575
- [Background] de Jong Z, Munneke M, Zwinderman AH, Kroon HM, Jansen A, Ronday KH, van Schaardenburg D, Dijkmans BA, Van den Ende CH, Breedveld FC, Vliet Vlieland TP, Hazes JM. Is a long-term high-intensity exercise program effective and safe in patients with rheumatoid arthritis? Results of a randomized controlled trial. Arthritis Rheum. 2003 Sep;48(9):2415-24. doi: 10.1002/art.11216. PMID 13130460
- [Background] van den Ende CH, Breedveld FC, le Cessie S, Dijkmans BA, de Mug AW, Hazes JM. Effect of intensive exercise on patients with active rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2000 Aug;59(8):615-21. doi: 10.1136/ard.59.8.615. PMID 10913058